CLINICAL TRIAL: NCT03605771
Title: Descriptive Observational Study on the Characteristics of Advanced and Metastatic Melanoma in Spain
Acronym: GEM-1801
Status: Recruiting | Type: Observational
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Responsible Party: Sponsor
Other Study IDs: GEM-1801
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Melanoma Stage Iv; Melanoma Stage Iii; Advanced Cancer
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Advanced Melanoma: Patients of legal age with stage III, metastatic, or unresectable melanoma at first diagnosis after January 8, 2018. First diagnosis is understood as:
  1. Disease onset as metastatic or unresectable disease.
  2. First metastatic or unresectable relapse in the pre-established dates (after January 8, 2018) in a patient with previous localised melanoma and completely resected on dates before the pre-inclusion period.
  Interventions: Other: Daily Clinical Practice

INTERVENTIONS:
Other: Daily Clinical Practice — The assignment of a patient to a specific therapeutic strategy will not be decided in advance by the study protocol, but will be determined by the usual clinical practice of medicine, and the decision to prescribe a specific treatment will be clearly dissociated from the decision to include a patient in the study. No intervention will be applied to patients, either diagnostic or follow-up, other than the usual clinical practice.

SUMMARY:
This is an observational, multicentre epidemiological study with a longitudinal cohort in which information will be retrieved from medical records of patients with advanced metastatic or unresectable melanoma at first diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age with stage III, metastatic, or unresectable melanoma at first diagnosis after January 8, 2018. First diagnosis is understood as: a. Disease onset as metastatic or unresectable disease; b. First metastatic or unresectable relapse in the pre-established dates (after January 8, 2018) in a patient with previous localised melanoma and completely resected on dates before the pre-inclusion period.
* Signing the Informed Consent Form (ICF).
* A patient may have received the first or subsequent treatments for metastatic or unresectable disease in a hospital other than the centre where the ICF was signed, as long as the patient meets the inclusion criteria 1.
* A patient can only sign one ICF (cannot sign an ICF in two different centres).
* If a patient signs the ICF in a centre during the first-line therapy and then goes to another centre with consideration for the following lines: If the centre is associated with the GEM-1801 study, researchers will do their best to update the following lines and the patient status, introducing the new information in the centre where the ICF was initially signed. This information will be provided by the patient before contacting the principal investigator and always with prior consent of the patient, who will have previously provided the consent to contact by telephone for this purpose. If this second (or subsequent) centre is not associated with the GEM- 1801 study, this will be considered loss of follow-up, unless the patient returns to the GEM-1801 start centre, wherein the reporting physicians will do their best to update the information from other centres, always with prior patient consent, who will have previously signed the ICF; c) A patient card with the assigned code will be delivered.

Exclusion Criteria:

* Any patient not complying with inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A 'case' is defined as any patient, diagnosed, treated, or followed in the different health centres where reporting physicians authorised by the GEM group work, who meets the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sample Characteristics | Baseline
  Sociodemographic and disease characteristics of patients diagnosed with stage III, metastatic or unresectable melanoma at first diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Iván Márquez Rodas, M.D., Study Chair — Hospital General Universitario Gregorio Marañón; Salvador Martín Algarra, M.D., Principal Investigator — Clínica Universidad de Navarra
Locations (39):
- Spain (39):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Onconogranada, Granada, Andalusia
  - Hospital Universitario Regional de Málaga, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Araba Txagorritxu Victoria, Vitoria-Gasteiz, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitario Río Hortega, Valladolid, Castille and León
  - Hospital General de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Instituto Catalán de Oncología Badalona, Badalona, Catalonia
  - Hospital de la Santa Creu y Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Quirón Dexeus, Barcelona, Catalonia
  - Hospital Universitario San Pedro Alcántara, Cáceres, Extremadura
  - Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Lucus Augusti, Lugo, Lugo
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Son Llàtzer, Palma de Mallorca, Palma
  - Complejo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Hospital Universitario de Valme, Seville, Sevilla
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Hospital La Ribera, Alzira, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cerezuela-Fuentes P, Pinero-Madrona A, Munoz-Couselo E, Manzano JL, Berciano-Guerrero MA, Majem M, Espinosa E, Soria A, Ayala de Miguel P, Garcia Castano A, Crespo G, Gutierrez Sanz L, Aguado de la Rosa C, Fernandez-Morales LA, Puertolas T, Fra Rodriguez J, Rodriguez de la Borbolla M, Bellido L, Lopez Castro R, Navarro Perez V, Garcia Arroyo FR, Villa Guzman JC, Campos Balea B, Hernandez B, Martin Algarra S, Marquez-Rodas I. Title: Characterization of Melanoma of Unknown Primary in the Era of Immunotherapy and Targeted Therapy in Spain: Results from the Prospective Real World Study GEM 1801. Clin Transl Oncol. 2025 Dec 20. doi: 10.1007/s12094-025-04164-w. Online ahead of print. PMID 41420791
- [Derived] Espinosa E, Berciano-Guerrero MA, Munoz-Couselo E, Puertolas T, Manzano JL, Soria A, de Miguel PA, Crespo G, Sanz LG, Cerezuela-Fuentes P, de la Rosa CA, Majem M, Castano AG, Berrocal A, Arroyo FRG, de la Borbolla MR, Bellido L, Martinez JM, Fernandez LA, Carnicero AM, Castro RL, Rodriguez AB, Lecumberri MJ, Guzman JCV, Balea BC, Rodriguez JF, Bautista JV, Perez VN, Mujika K, Subias MC, Hernandez B, Algarra SM, Marquez-Rodas I. Response rate and long-term survival in patients with advanced melanoma: data from the prospective cohort study gem-1801. Clin Transl Oncol. 2025 Nov 28. doi: 10.1007/s12094-025-04098-3. Online ahead of print. PMID 41313559
- [Derived] Ayala-de Miguel P, Munoz-Couselo E, Gutierrez-Sanz L, Fernandez LA, Navarro-Perez V, Berciano-Guerrero MA, Garcia-Arroyo F, Aguado-de la Rosa C, Cerezuela-Fuentes P, Majem M, Campos-Balea B, Soria A, Hernandez-Marin B, Garcia-Castano A, Martin-Algarra S, Marquez-Rodas I. Retreatment and rechallenge with BRAF/MEK inhibitors in patients with metastatic melanoma: results from the real-world Spanish Melanoma Registry (GEM-1801). Clin Transl Oncol. 2026 Jan;28(1):320-329. doi: 10.1007/s12094-025-04005-w. Epub 2025 Jul 27. PMID 40715648